CLINICAL TRIAL: NCT05538897
Title: A Phase IB and Randomized Phase II Trial of Megestrol Acetate With or Without Ipatasertib in Recurrent or Metastatic Endometrioid Endometrial Cancer
Brief Title: Testing the Addition of the AKT Inhibitor, Ipatasertib, to Treatment With the Hormonal Agent Megestrol Acetate for Recurrent or Metastatic Endometrial Cancers
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2022-07505; NCI-2022-07505 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-GY028 (Other: NRG Oncology); NRG-GY028 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2022-09-13; First posted 2022-09-14 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: FIGO Grade 1 Endometrial Endometrioid Adenocarcinoma; FIGO Grade 2 Endometrial Endometrioid Adenocarcinoma; Metastatic Endometrial Endometrioid Adenocarcinoma; Recurrent Endometrial Endometrioid Adenocarcinoma
MeSH Terms: interventions — Specimen Handling; ipatasertib; Magnetic Resonance Spectroscopy; Megestrol Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Phase Ib (megestrol acetate, ipatasertib) (Experimental): Patients receive megestrol acetate PO QD on days 1-28 and ipatasertib PO QD on days 1-21 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo a CT or MRI during screening, on study, and during follow-up. Patients also undergo collection of blood samples throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Ipatasertib; Procedure: Magnetic Resonance Imaging; Drug: Megestrol Acetate
- Phase II (megestrol acetate) (Active Comparator): Arm I: Patients receive megestrol acetate PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo a CT or MRI during screening, on study, and during follow-up. Patients also undergo collection of blood samples throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Megestrol Acetate
- Phase II (megestrol acetate, ipatasertib) (Experimental): Arm II: Patients receive megestrol acetate PO QD on days 1-28 and ipatasertib PO QD on days 1-21 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo a CT or MRI during screening, on study, and during follow-up. Patients also undergo collection of blood samples throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Ipatasertib; Procedure: Magnetic Resonance Imaging; Drug: Megestrol Acetate

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Ipatasertib — Given PO
  Other Names: GDC 0068; GDC-0068; GDC0068; RG 7440; RG-7440; RG7440
  Arms: Phase II (megestrol acetate, ipatasertib); Phase Ib (megestrol acetate, ipatasertib)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Megestrol Acetate — Given PO
  Other Names: 17-Hydroxy-6-methylpregna-4,6-diene-3,20-dione acetate; 17.alpha.-Acetoxy-6-methylpregna-4,6-diene-3,20-dione; 6-Dehydro-6-methyl-17.alpha.-acetoxyprogesterone; 6-Methyl-6-dehydro-17.alpha.-acetoxyprogesterone; BDH 1298; BDH-1298; Maygace; Megace; Megestat; Megestil; Niagestin; Ovaban; Pallace; SC 10363; SC-10363

SUMMARY:
This phase Ib/II trial tests the safety, side effects, best dose, and effectiveness of the combination of ipatasertib with megestrol acetate to megestrol acetate alone in patients with endometrial cancer that has come back (recurrent) or has spread to other places in the body (metastatic). Ipatasertib may stop the growth of tumor cells and may kill them by blocking some of the enzymes needed for cell growth. Megestrol acetate lowers the amount of estrogen and also blocks the use of estrogen made by the body. This may help stop the growth of tumor cells that need estrogen to grow. The combination of ipatasertib and megestrol acetate may be more effective in treating endometrial cancer than megestrol acetate alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the toxicity of ipatasertib in combination with megestrol acetate in women with metastatic grade 1-2 endometrioid endometrial cancer and establish the recommended phase II dose. (Phase I) II. Compare the progression free survival of the combination of ipatasertib with megestrol acetate to megestrol acetate alone among women with metastatic grade 1-2 endometrioid adenocarcinoma of the endometrium. (Phase II) III. Compare the toxicity of the combination of ipatasertib with megestrol acetate to megestrol acetate alone. (Phase II)

SECONDARY OBJECTIVES:

I. Compare objective response rate per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 between the two arms.

II. Examine the pharmacokinetics of ipatasertib + megestrol acetate to assess potential drug-drug interactions.

III. Assess the association between biomarkers and response to therapy.

EXPLORATORY OBJECTIVE:

I. Explore whether pS6/total S6 and pPRAS40/total PRAS40 expression is impacted by the use of ipatasertib and megestrol acetate.

OUTLINE: This is a phase Ib, dose de-escalation study of ipatasertib followed by a phase II study.

PHASE Ib: Patients receive megestrol acetate orally (PO) once daily (QD) on days 1-28 and ipatasertib PO QD on days 1-21 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo a computed tomography (CT) or magnetic resonance imaging (MRI) during screening, on study, and during follow-up. Patients also undergo collection of blood samples throughout the trial.

PHASE II: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive megestrol acetate PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo a CT or MRI during screening, on study, and during follow-up. Patients also undergo collection of blood samples throughout the trial.

ARM II: Patients receive megestrol acetate PO QD on days 1-28 and ipatasertib PO QD on days 1-21 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo a CT or MRI during screening, on study, and during follow-up. Patients also undergo collection of blood samples throughout the trial.

After completion of study treatment, patients are followed up at 30 days for the phase I study. Patients are followed up every 3 months for 2 years, then every 6 months for 3 years for the phase II study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have grade 1 or 2 recurrent or metastatic endometrioid endometrial cancer
* Patients must have measurable disease according to RECIST version (v)1.1. Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded). Each lesion must be >= 10 mm when measured by CT or MRI. Lymph nodes must be >= 15 mm in short axis when measured by CT or MRI. Previously irradiated lesions can be considered as measurable disease only if progressive disease has been unequivocally documented at that site since radiation
* Patients may have received unlimited prior lines of therapy. If patient received prior hormonal therapy (e.g., megestrol acetate, medroxyprogesterone acetate, aromatase inhibitor, tamoxifen, fulvestrant) it must have completed at least 6 months prior to registration
* Age >= 18
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1 or 2
* Platelets >= 100,000/mcl within 14 days prior to registration
* Absolute neutrophil count (ANC) >= 1,500/mcl within 14 days prior to registration
* Hemoglobin >= 9 g/dL within 14 days prior to registration
* Glomerular filtration rate (GFR) >= 60 mL/min/1.73m^2 measured using Cockcroft-Gault equation or the estimated glomerular filtration rate from the Modification of Diet in Renal Disease Study within 14 days prior to registration
* Total bilirubin =< 1.5 x the upper limit of normal (ULN) within 14 days prior to registration

  * Patients with known Gilbert syndrome who have bilirubin =< 3 x ULN may be enrolled
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional ULN within 14 days prior to registration
* Albumin >= 3 g/dL within 14 days prior to registration
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* The effects of ipatasertib on the developing human fetus are unknown. For this reason and because AKT inhibitor agents as well as other therapeutic agents used in this trial are known to be teratogenic, participants of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) during study therapy and for 28 days following the last dose of study therapy. Should a participant become pregnant or suspect pregnancy while participating in this study, they should inform their treating physician immediately
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* For patients with known human immunodeficiency virus (HIV), hepatitis B virus (HBV), and/or hepatitis C virus (HCV) infection:

  * HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months of registration are eligible for this trial
  * Patients with evidence of chronic hepatitis B virus (HBV) infection must have an undetectable HBV viral load on suppressive therapy, if indicated
  * Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression
* Patients must be able to swallow and retain oral medications and not have gastrointestinal illnesses that would preclude absorption of megestrol acetate or ipatasertib as judged by the treating physician
* The patient or a legally authorized representative must provide study-specific informed consent prior to study entry and, for patients treated in the United States (U.S.), authorization permitting release of personal health information

Exclusion Criteria:

* Patients who have had prior treatment with an AKT inhibitor (Prior treatment with PI3K or mTOR inhibitors is allowed)
* Patients who have received treatment with strong CYP3A inhibitors or inducers within 14 days or 5 drug-elimination half-lives, whichever is longer, prior to study registration

  * Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Patients with diabetes either requiring insulin therapy or with a baseline fasting glucose > 160 mg/dL and/or high glycosylated hemoglobin A1c (HbA1c) (> 8), suggesting poorly controlled diabetes. Fasting is defined as abstaining from food and drink (with the exception of water) for at least 8 hours
* Patients who require chronic corticosteroid therapy of > 10 mg of prednisone per day or an equivalent dose of other anti-inflammatory corticosteroids or immunosuppressant agents for a chronic disease
* Patients with grade 2 or greater uncontrolled or untreated hypercholesterolemia (> 300 mg/dL) or hypertriglyceridemia (> 300 mg/dL)
* Patients with a history of known or active inflammatory bowel disease (e.g., Crohn disease and ulcerative colitis) or active bowel inflammation (e.g., diverticulitis)
* Patients with a history of or presence of an abnormal electrocardiogram (ECG) that is clinically significant in the investigator's opinion (including complete left bundle branch block, second- or third-degree heart block, or evidence of prior myocardial infarction)
* Patients with known clinically significant history of liver disease consistent with Child-Pugh class B or C, including active viral or other hepatitis, current drug or alcohol abuse, or cirrhosis
* Patients with lung disease: Grade 2 or greater pneumonitis, grade 2 or greater interstitial lung disease, idiopathic pulmonary fibrosis, cystic fibrosis, aspergillosis, active tuberculosis, or history of opportunistic infections (pneumocystis pneumonia or cytomegalovirus pneumonia) within the past 6 months
* No active infection requiring parenteral antibiotics
* Women who are pregnant or unwilling to discontinue nursing

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-03-31 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) (Phase Ib) | Up to 5 years
  To determine frequency and severity of adverse events for all dose combinations of megestrol acetate plus ipatasertib. Descriptive statistics will be used to summarize AEs. These analyses will focus on individuals who initiated their assigned treatment and will summarize maximum grade of AEs occurring during treatment classified by Common Toxicity Criteria (CTC) category. The primary summary of AEs will present counts and percentages, regardless of whether the AE was attributed to any of the study agents.
Maximum tolerated dose for phase II (Phase Ib) | Up to 5 years
  Descriptive statistics will be used to summarize AEs. These analyses will focus on individuals who initiated their assigned treatment and will summarize maximum grade of AEs occurring during treatment classified by CTC category. The primary summary of AEs will present counts and percentages, regardless of whether the AE was attributed to any of the study agents.
Progression free survival (PFS) (Phase II) | From study entry to time of progression or death, whichever occurs first, or date of last contact if neither progression nor death has occurred, assessed up to 5 years
  Compare PFS of the combination of ipatasertib with megestrol acetate to megestrol acetate alone among women with recurrent/metastatic endometrioid adenocarcinoma of the endometrium. A product-limit method will be used to estimate the cumulative distribution of PFS duration for each of the study treatments used in this population.
Incidence of AEs (Phase II) | Up to 5 years
  Summarize the toxicity/adverse events of the combination of ipatasertib with megestrol acetate and megestrol acetate alone. Adverse events will be categorized using Common Terminology Criteria for Adverse Events version 5.0.

SECONDARY OUTCOMES:
Pharmacokinetics of ipatasertib + megestrol acetate (Phase Ib) | On cycle 1, day 8
  Examine the pharmacokinetics of ipatasertib + megestrol acetate to assess potential drug-drug interactions. This data will be summarized descriptively.
Objective response rate (Phase II) | Up to 5 years
  Response is defined as complete response or partial response (CR+PR) evaluated by Response Evaluation Criteria in Solid Tumors version 1.1. A logistic model will be used to estimate the relative odds of responding (CR+PR) to megestrol acetate + ipatasertib relative to megestrol acetate alone after adjusting for prior progesterone therapy.
Biomarkers (Phase II) | Up to 5 years
  The association between biomarkers and response to therapy will be assessed. Integrated biomarker endpoints include: PTEN immunohistochemistry, estrogen receptor and progesterone receptor, whole exome sequencing, ribonucleic acid sequencing. Proportional hazards models will be used to examine the prognostic association of integrated biomarkers with PFS; and interactions between markers and treatment arm will be used to examine the markers' predictive association with PFS.

OTHER OUTCOMES:
pS6/total S6 and pPRAS40/total PRAS40 expression (Phase II) | Up to 5 years
  Exploratory objectives include assessing whether pS6/total S6 and pPRAS40/total PRAS40 expression is impacted by the use of ipatasertib and megestrol acetate. Exploratory biomarker results will be provided to the NRG Oncology Statistical and Data Management Center for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Michaela O Grinsfelder, Principal Investigator — NRG Oncology
Locations (152):
- United States (152):
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Highlands Oncology Group - Fayetteville, Fayetteville, Arkansas
  - Highlands Oncology Group - Rogers, Rogers, Arkansas
  - Highlands Oncology Group, Springdale, Arkansas
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Sarasota Memorial Hospital-Venice, N. Venice, Florida
  - Florida Cancer Specialists - Sarasota Downtown, Sarasota, Florida
  - First Physicians Group-Sarasota, Sarasota, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Florida Cancer Specialists - Venice Pinebrook, Venice, Florida
  - Augusta University Medical Center, Augusta, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Northwestern University, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Northwestern Medicine Grayslake Outpatient Center, Grayslake, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - IU Health North Hospital, Carmel, Indiana
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - Goshen Center for Cancer Care, Goshen, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo Cancer Center, Kalamazoo, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Community Medical Center, Missoula, Montana
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - Summa Health System - Akron Campus, Akron, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Miami Valley Cancer Care and Infusion, Greenville, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - UH Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Jefferson Hospital, Jefferson Hills, Pennsylvania
  - Forbes Hospital, Monroeville, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - Wexford Health and Wellness Pavilion, Wexford, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Memorial Hermann Texas Medical Center, Houston, Texas
  - UT Southwestern Clinical Center at Richardson/Plano, Richardson, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Carilion Roanoke Memorial Hospital, Roanoke, Virginia
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

DOCUMENTS (2):
  • Informed Consent Form: Phase I consent (2025-01-03): https://cdn.clinicaltrials.gov/large-docs/97/NCT05538897/ICF_000.pdf
  • Informed Consent Form: Phase II consent (2025-01-03): https://cdn.clinicaltrials.gov/large-docs/97/NCT05538897/ICF_001.pdf